CLINICAL TRIAL: NCT05216289
Title: The Efficacy of an Oral Probiotic Associated With a Fixed Combination of Benzoyl Peroxide and Adapalene in the Treatment of Acne: A Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: The Efficacy of an Oral Probiotic Associated With a Fixed Combination of Benzoyl Peroxide and Adapalene in the Treatment of Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Medcin Instituto da Pele Ltda (Unknown)
Responsible Party: Principal Investigator, Marco Alexandre Dias da Rocha, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Probiac
Record Dates: First submitted 2021-12-19; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Acne Vulgaris
Keywords: probiotic; acne; adapalene; benzoyl peroxide; microbiome
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- probiac + topical fixed combination (Active Comparator)
  Interventions: Dietary Supplement: Probiac
- placebo + topical fixed combination (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiac — Oral probiotic composed of Lactobacillus acidophilus, Bifidobacterium lactis, vitamins and minerals - Exímia Probiac® (EP), in combination with 2.5% benzoyl peroxide plus 0.1% adapalene (PBA) for topical use.
  Arms: probiac + topical fixed combination
Other: Placebo — Placebo + 2.5% benzoyl peroxide plus 0.1% adapalene (PBA) for topical use.
  Arms: placebo + topical fixed combination

SUMMARY:
Objective: Clinical trial carried out to evaluate the superiority of efficacy of a treatment regimen with an oral probiotic associated with a fixed combination of 0.1% adapalene and 2.5% benzoyl peroxide compared to an oral placebo with the same topical treatment in patients with mild to moderate acne.

Patients and Methods: This was a randomized, double-blind, placebo-controlled study conducted with 212 patients aged from 12 to 35 years; 107 in the test treatment arm and 105 in the comparator arm. The study was divided into two phases of 90 days each, totaling 180 days. In the first phase, patients received treatment with 2.5% benzoyl peroxide and 0.1% adapalene associated with a probiotic (IT), or 2.5% benzoyl peroxide and 0.1% adapalene associated with placebo (CT). In the second phase (90 days), patients received only oral treatment with a probiotic or placebo. Efficacy criteria were: reduction of the Investigator Global Assessment (IGA) scale to 0 or 1, and reduced lesion count.

DETAILED DESCRIPTION:
Four hundred participants of both genders aged between 12 and 35 years, diagnosed with grade II and III acne, mixed or oily skin and phototype between I and IV, according to the Fitzpatrick scale, were recruited. Pregnant or lactating women, as well as those intending to become pregnant during the study period were excluded, in addition to patients who received treatment with corticosteroids and antimicrobials within 30 days prior to selection and those who were treated with immunosuppressants within 90 days prior to selection.

The study was conducted in Osasco-SP, Brazil, at Medcin Instituto da Pele Ltda., in the period from April 18th, 2018 to April 7th, 2021. The study protocol was approved by the Research Ethics Committee at Universidade São Francisco-SP on December 14, 2018. CAAE: 03728318.5.0000.5514 Opinion Number: 3,083,043. All participants signed the Informed Consent Form (ICF) and the research was conducted in accordance with Good Clinical Practice and the 1996 Declaration of Helsinki.

Study Design and Treatment This was a randomized, double-blind, 2-arm, placebo-controlled study conducted to assess the superiority of treatment with the oral probiotic composed of Lactobacillus acidophilus, Bifidobacterium lactis, vitamins and minerals - Exímia Probiac® (EP), in combination with 2.5% benzoyl peroxide plus 0.1% adapalene (PBA) for topical use, compared to PBA in combination with placebo in improving the clinical condition of acne patients.

Eligible patients were randomized into 2 groups to receive one of the treatments. Both topical and oral treatments were administered once a day. All patients received a bottle of SPF50 sunscreen on the first visit and were instructed to use it daily. All study samples were supplied by the company Farmoquímica S/A.

The study was divided into two phases of 90 days each, totaling 180 days of study. Patients were evaluated at the baseline visit (D0) and every 30 days thereafter, totaling 7 visits. At Day 0 visit, patients received the randomized treatment and guidelines for use. In the first phase (90 days), patients received treatment with PBA plus PE (Investigational Treatment - IT) or PE plus placebo (Comparator Treatment - CT). In the second phase (90 days), patients received only oral treatment with PE or placebo.

At each visit (Day 0, Day 30, Day 60, Day 90, Day 120, Day 150 and Day 180), patients were clinically evaluated and the results in relation to the Investigator Global Assessment (IGA) scale were recorded.

Efficacy criteria

The primary variables of the study were the reduction in the IGA scale score to grade 1 or 0, as well as the reduction in the total number of inflammatory and non-inflammatory lesions in the facial region. For IGA quantification, scores were assigned according to an established scale:

0 = Clean skin: Residual hyperpigmentation and erythema may be present;

1. = Almost clean: Some scattered comedones and some small papules;
2. = Mild: Less than half of the face is affected, some comedones and some papules and pustules;
3. = Moderate: More than half of the face is affected, some comedones and some papules and pustules. A lump may be present;
4. = Severe: Whole face severely affected by comedones, numerous papules and pustules, and some nodules and cysts.

Statistical analysis

The results obtained from clinical, instrumental and subjective evaluations were compared between experimental time points and later between treatments. The hypothesis tests used in the study had a significance level of 95% and the statistical power of these tests was above 80%. Descriptive analyses of the study variables were performed using frequency tables and descriptive statistics. The percentage of participants with a reduction in the total number of inflammatory and non-inflammatory lesions, the percentage of participants with regression of the IGA scale score to no lesions (score zero) or almost no lesions (score one) were evaluated using the Z test for comparison of two proportions. The results were considered statistically significant at a significance level of 5% (p-value ≤0.05). The significance level was controlled by rejecting the null hypotheses if the p-value was less than or equal to 5%.

ELIGIBILITY:
Inclusion Criteria:

participants of both genders aged between 12 and 35 years, acne grade II and III acne mixed or oily skin phototype between I and IV, according to the Fitzpatrick scale, were recruited

Exclusion Criteria:

Pregnant or lactating women, as well as those intending to become pregnant during the study period patients who received treatment with corticosteroids and antimicrobials within 30 days prior to selection patients who were treated with immunosuppressants within 90 days prior to selection.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment (IGA) | day 30
  patients were clinically evaluated and the results in relation to the Investigator Global Assessment (IGA)
Investigator Global Assessment (IGA) | day 60
  patients were clinically evaluated and the results in relation to the Investigator Global Assessment (IGA)
Investigator Global Assessment (IGA) | day 90
  patients were clinically evaluated and the results in relation to the Investigator Global Assessment (IGA)
Investigator Global Assessment (IGA) | day 120
  patients were clinically evaluated and the results in relation to the Investigator Global Assessment (IGA)
Investigator Global Assessment (IGA) | day 150
  patients were clinically evaluated and the results in relation to the Investigator Global Assessment (IGA)
Investigator Global Assessment (IGA) | day 180
  patients were clinically evaluated and the results in relation to the Investigator Global Assessment (IGA)

SECONDARY OUTCOMES:
Lesion | day 30
  number of inflammatory and non inflammatory lesions
Lesion | day 60
  number of inflammatory and non inflammatory lesions
Lesion | day 90
  number of inflammatory and non inflammatory lesions
Lesion | day 120
  number of inflammatory and non inflammatory lesions
Lesion | day 150
  number of inflammatory and non inflammatory lesions
Lesion | day 180
  number of inflammatory and non inflammatory lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele Ltda, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT05216289/SAP_000.pdf
  • Informed Consent Form (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT05216289/ICF_001.pdf